CLINICAL TRIAL: NCT01141049
Title: Gabapentin for Abstinence Initiation in Alcohol Dependence
Acronym: GAINS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, John Mariani MD, research psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #6123
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Results first posted 2018-07-18 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Alcohol Dependence
Keywords: Alcohol Withdrawal; Reducing Alcohol Consumption; Promoting abstinence in alcohol-dependent patients; Gabapentin
MeSH Terms: conditions — Alcoholism | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin (Active Comparator): Gabapentin will be titrated over a 7-day period to the dose target or the maximum tolerated dose. The maximum dose will be 1200mg TID. Participants must be able to tolerate and comply with at least 400 mg daily.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Placebo capsules will be administered TID.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gabapentin — During week 1 the dosage will be increased 3 times. Days 1 and 2, participants will receive 400 mg of Gabapentin three times daily. During days 3 and 4 the dosage will be increased to 800 mg three times daily. On day 5 through 7, participants will receive a dose of 1200 mg three times daily, which will continue from week 2 through 8. During week 9 patients will be tapered off for the duration of the week.
  Other Names: Neurontin
  Arms: Gabapentin
Other: Placebo — Placebo, TID
  Arms: Placebo

SUMMARY:
Primary Hypotheses:

1. Gabapentin will significantly reduce alcohol consumption and promote abstinence as compared to placebo. The primary outcome measure will be the number of the heavy drinking days (defined as any day where the number of standard drinks was at least 5 for men and at least 4 for women) per week as measured by the timeline follow-back method.

Secondary Hypotheses:

1. Gabapentin will be superior to placebo in reducing alcohol use as measured by percent days abstinent.

DETAILED DESCRIPTION:
In an 8-week randomized double-blind placebo-controlled outpatient pilot trial the efficacy of gabapentin in the treatment of alcohol dependence will be studied in 60 patients. Participants will be randomly assigned to treatment under double-blind conditions with either 1) a fixed dosing schedule of gabapentin or 2) placebo. All participants will receive weekly supportive behavioral treatment that promotes abstinence from alcohol and other substances, encourages mutual-support meeting attendance, and facilitates compliance with study medication. The primary outcome measures will be: the reduction of heavy drinking days per week as measured by the timeline follow-back method.

Participants will be alcohol-dependent men and nonpregnant women who report drinking a minimum of 5 standard drinks for men or 4 standard drinks for women at least 4 days per week over the past 28 days. The daily minimum drinking requirements are consistent with the commonly accepted definition of "binge drinking." A minimum requirement of having a heavy drinking episode 4 days a week would select for a population of individuals who are drinking excessively more days than not. A minimum threshold of weekly alcohol use is set to prevent a "floor effect" (i.e. participants with minimal alcohol use at baseline would be unable to demonstrate significant improvement.)

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65.
* Meets DSM-IV criteria for current alcohol dependence.
* Seeking treatment for alcohol dependence.
* Reports drinking a minimum of 5 standard drinks for men or 4 standard drinks for women at least 4 days per week over the past 28 days.
* Able to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Lifetime history of DSM-IV diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder.
* A diagnosis of current major depressive disorder or any other current Axis I psychiatric disorder as defined by DSM-IV-TR, other than alcohol dependence, that in the investigator's judgment might require intervention with either pharmacological or non-pharmacological therapy over the course of the study.
* Patients currently taking prescribed psychotropic medications that would be disrupted by study medication or by an effort to discontinue alcohol use.
* Evidence of moderate-to-severe alcohol withdrawal (CIWA-Ar > 13.
* History of allergic reaction to candidate medication (gabapentin).
* History of alcohol withdrawal seizures or alcohol withdrawal delirium.
* Pregnancy, lactation, or failure to use adequate contraceptive methods in female patients who are currently engaging in sexual activity with men.
* Unstable medical conditions, such as poorly controlled diabetes or hypertension (> 140/90 mm Hg), which might make participation hazardous.
* Subjects who have a current DSM-IV-TR diagnosis of other substance dependence, with the exception of nicotine and caffeine dependence. A diagnosis of substance abuse will not be exclusionary unless significant illicit substance use is present.
* Are legally mandated to participate in an alcohol use disorder treatment program.
* Who by history and current assessment represent a significant risk for suicide.
* Subjects who are likely, based on history, to place themselves in danger (e.g., driving while intoxicated or otherwise being unwilling to follow safety precautions).
* Renal insufficiency or abnormal renal function.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mariani, MD, Principal Investigator — NYSPI
Locations (2):
- United States (2):
  - Substance Treatment and Research Service (STARS), New York, New York
  - New York State Psychiatric Institute, New York, New York

REFERENCES:
- [Derived] Mariani JJ, Pavlicova M, Basaraba C, Mamczur-Fuller A, Brooks DJ, Bisaga A, Carpenter KM, Nunes EV, Levin FR. Pilot randomized placebo-controlled clinical trial of high-dose gabapentin for alcohol use disorder. Alcohol Clin Exp Res. 2021 Aug;45(8):1639-1652. doi: 10.1111/acer.14648. Epub 2021 Jul 5. PMID 34120336

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 19 | 21
Completed | 14 | 13
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (9.5) | 49.8 (8.7) | 48.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 11 | 11 | 22
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent of Heavy Drinking Days Per Week
Description: percent of heavy drinking days as defined as 5 drinks per day for males and 4 drinks per day for females over the course of a study week.
Time Frame: assesed over 8 weeks, presented for week 8 of trial
Measure: Mean (Standard Deviation); unit: percent of heavy drinking days
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 19 | 21
percent of heavy drinking days | 22.5 (34.0) | 53.9 (44.0)

2. Secondary Outcome: Percent Days of Abstinence From Alcohol
Description: During the course of 8 weeks the medication aims to determine whether it is effective in reducing alcohol consumption, and promoting abstinence in alcohol-dependent patients.
Time Frame: assessed for up to 8 weeks, presented at week 8 of trial
Measure: Mean (Standard Deviation); unit: percent of days abstinent
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 19 | 21
percent of days abstinent | 50 (37) | 27.5 (38)

ADVERSE EVENTS:
Time Frame: during 8 weeks of trial or participant's length of participation
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 15/19 | 11/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=19) | Placebo (N=21)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
anxiety (General disorders) | 0 (0) | 1 (1)
appetite change (Gastrointestinal disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
dizziness (General disorders) | 2 (2) | 1 (1)
dry mouth (General disorders) | 3 (3) | 4 (4)
headache (General disorders) | 2 (2) | 2 (2)
gi upset (Gastrointestinal disorders) | 0 (0) | 1 (1)
insomnia (General disorders) | 1 (1) | 0 (0)
libido changes (General disorders) | 0 (0) | 1 (1)
muscle pain/weakness (General disorders) | 0 (0) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
somnolence (General disorders) | 2 (2) | 1 (1)
fatigue (General disorders) | 2 (2) | 5 (5)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes